CLINICAL TRIAL: NCT07382375
Title: AI-assisted Immunoinflammatory Subtyping-Directed Precision Treatment in Acute Aortic Dissection: A Multicenter RCT-based Exploration
Brief Title: AI-assisted Subtyping-directed Precision Treatment in Acute Aortic Dissection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Third Affiliated Hospital of Soochow University (Unknown); West China Hospital (Other); Fujian Medical University Union Hospital (Other); Shanghai East Hospital (Other); Beijing Anzhen Hospital (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PANDA-Smart
Record Dates: First submitted 2026-01-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Aortic Aneurysm and Dissection
Keywords: inflammation; immune
MeSH Terms: conditions — Aortic Dissection; Inflammation | interventions — urinastatin; Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subtyping-based precision therapy (Experimental): * Balanced type (HIS1): No anti-inflammatory intervention required;
    * Inflammation-excessive type (HIS2): Anti-inflammatory intervention with ulinastatin; ③ Immunosuppressive type (HIS3): Immunomodulation with thymalfasin; ④ Mixed reaction type (HIS4): Combined treatment with ulinastatin and thymalfasin.
  Interventions: Drug: Ulinastatin and Thymalfasin
- Conventional Empirical Strategy (Active Comparator): treatment of physician's choice alone
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin and Thymalfasin — AI-assisted Immunoinflammatory Subtyping-guided Target-matching Individualized Anti-inflammatory Strategy
  Arms: Subtyping-based precision therapy
Drug: Ulinastatin — Conventional empirical regimens will be formulated based on patients' clinical symptoms and routine inflammatory indicators (white blood cell count, C-reactive protein, procalcitonin) without uniform target-matching standards, with reference to clinical diagnosis and treatment guidelines: if obvious inflammatory responses are present (e.g., fever, significant elevation of C-reactive protein), non-steroidal anti-inflammatory drugs or low-dose glucocorticoids will be administered; if complicated with infection, combined antibiotic therapy will be given; for patients with normal or slightly elevated inflammatory indicators, anti-inflammatory drugs may be temporarily withheld, and close monitoring will be performed instead. The regimen will be adjusted according to changes in routine inflammatory indicators after surgery until the patient is discharged.
  Arms: Conventional Empirical Strategy

SUMMARY:
Aortic dissection has acute onset and high mortality, with immunoinflammatory response driving lesion progression. Current perioperative anti-inflammatory therapies are mostly empirical and poorly targeted, and AI-assisted typing lacks a complete clinical translation pathway. This study integrates multi-dimensional data to construct an AI immunoinflammatory subtyping system, enabling rapid subtyping and establishing a "subtyping-target-treatment" closed loop for emergency needs. Using a prospective multicenter RCT, 300 patients are randomly divided into two groups: the experimental group receives subtyping-based precision therapy, while the control group uses empirical strategies (treatment of physician's choice). It observes 7-day postoperative SOFA score, SIRS and other prognostic indicators to provide evidence-based support for precision treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of acute aortic dissection by contrast-enhanced Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA);
2. Planned emergency surgical treatment (including open surgery and endovascular repair);
3. Aged 18-80 years old, regardless of gender;
4. Time from onset to hospital admission ≤ 72 hours;
5. Signed informed consent form by the patient or their authorized agent, with willingness to cooperate with the follow-up of the study.

Exclusion Criteria:

1. Complicated with underlying diseases that affect immunoinflammatory status, such as severe infections (e.g., sepsis, infective endocarditis), autoimmune diseases, malignant tumors, chronic liver diseases, and chronic kidney diseases (uremic stage);
2. Long-term use of immunosuppressants or glucocorticoids before surgery (continuous use for ≥ 2 weeks);
3. Pregnant or lactating women;
4. Patients with mental disorders or cognitive dysfunction who cannot cooperate with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2027-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score. The SOFA score evaluates 6 organ systems, ranging from 0, no dysfunction, to 4, failure, and the total score ranges from 0, normal, to 24, most severe form of multiorgan failure. | 7 days after surgery
  The SOFA score evaluates 6 organ systems, ranging from 0, no dysfunction, to 4, failure, and the total score ranges from 0, normal, to 24, most severe form of multiorgan failure.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, Study Director — The First Affiliated Hospital with Nanjing Medical University; Hong Liu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (8):
- China (8):
  - Beijing Anzhen Hospital, Beijing
  - Changzhou First People Hospital, Changzhou
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Nanchang University Second Hospital, Nanchang
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Shanghai East Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No